CLINICAL TRIAL: NCT01511159
Title: A Single-Centre, Open-Label, Five-Period Crossover Trial In Healthy Male Volunteers Investigating the Relative Bioavailability of NNC 90-1170 By Pulmonary Administration Compared To A Subcutaneous Injection
Brief Title: Comparison of Liraglutide Inhaled Into the Lungs Compared to Liraglutide Injected Under the Skin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1464
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NNC 90-1170, initial dose (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Insulin (Active Comparator)
  Interventions: Drug: insulin human
- NNC 90-1170, final dose (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Single dose of 6 mcg/kg by inhalation. Progression to open-label trial part will be based on safety data
  Arms: NNC 90-1170, initial dose
Drug: placebo — Single dose by inhalation. Progression to open-label trial part will be based on safety data
  Arms: NNC 90-1170, initial dose
Drug: liraglutide — Single dose of 12 mcg/kg by inhalation. Subjects receive treatment in random order
  Arms: NNC 90-1170
Drug: liraglutide — Single dose 6 mcg/kg injected subcutaneously. Subjects receive treatment in random order
  Arms: NNC 90-1170
Drug: insulin human — Single dose 0.4 IU/kg by inhalation. Subjects receive treatment in random order
  Arms: Insulin
Drug: insulin human — Single dose 0.08 IU/kg injected subcutaneously. Subjects receive treatment in random order
  Arms: Insulin
Drug: liraglutide — 24 mcg/kg by inhalation. Progression to dose level will be based on safety evaluation
  Other Names: NNC 90-1170
  Arms: NNC 90-1170, final dose

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to determine the relative bioavailability of NNC 90-1170 (liraglutide) when inhaled compared to NNC 90-1170 when injected under the skin.

ELIGIBILITY:
Inclusion Criteria:

* No clinically important abnormal physical findings
* No clinically relevant abnormalities in the results of laboratory screening evaluation
* Normal (or abnormal but not clinically significant) ECG (electrocardiogram)
* Normal (or abnormal but not clinically significant) blood pressure and heart rate
* Body Mass Index (BMI) between 20-30 kg/m^2 or outwith range but not clinically significant
* Non-smoker
* Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1) at least 85% of predicted normal for age, gender and height
* FVC ratio at least 75% of predicted normal for age, gender and height

Exclusion Criteria:

* A clinically significant illness or infection requiring treatment within the last two months
* Any infection involving the respiratory system or adverse event that may, in the opinion of the principal investigator, interfere with blood glucose homeostasis
* Subjects with first and/or second degree relative(s) with diabetes mellitus
* Donation or loss of greater than 500 ml of blood in the period 0-12 weeks before trial entry
* Alcohol use in excess of 28 units of alcohol per week. A unit of alcohol is equivalent to half a pint of average strength beer, a glass (125 ml) of wine or a pub measure (25 ml) of spirits, sherry or port
* Current addiction to alcohol or substances of abuse
* Females
* Presence of hepatitis B surface antigen, hepatitis C antibody or HIV (human immunodeficiency virus) 1 or 2 antibodies

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2001-10; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Ratio of the areas under the plasma NN 90-1170 curves

SECONDARY OUTCOMES:
The maximum concentration (Cmax)
The time to maximum concentration (tmax)
Mean residence time (MRT)
Area under the curve
Terminal rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tranent, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com